CLINICAL TRIAL: NCT00322881
Title: A Phase II Study of Carboplatin and Paclitaxel in Elderly Women With Newly Diagnosed Ovarian, Peritoneal, or Fallopian Cancer
Brief Title: Carboplatin and Paclitaxel in Elderly Women With Newly Diagnosed Ovarian, Peritoneal, or Fallopian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early closure based on audit by study investigators after 3 patients died on study.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ursula A. Matulonis, MD, Medical Oncologist, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-402
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer; Mixed Tumor, Mesodermal
Keywords: carboplatin; paclitaxel; elderly women
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Mixed Tumor, Mesodermal | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin/Paclitaxel (Experimental): Patients received chemotherapy on day 1 of a 21 day cycle for 6 cycles. Paclitaxel was given via peripheral or central IV catheter at the dose of 175 mg/m2 over 3 hours. IV carboplatin followed using a dose of Area Under the Curve (AUC) equal to 5 with creatinine clearance based on Jelliffe formula.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Paclitaxel
  Other Names: Taxol
Drug: Carboplatin

SUMMARY:
The main purpose of this trial is to look at how elderly women (70 years of age or older) with newly diagnosed ovarian, peritoneal, or fallopian tube cancer manage six cycles of carboplatin and paclitaxel, what side effects they experience, and how their cancer reacts or responds to standard carboplatin and paclitaxel chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

•To determine the completion rate of six cycles of carboplatin/paclitaxel with no dose reductions because of toxicities.

Secondary

* Assess cancer antigen 125 (CA125) response rates of paclitaxel/carboplatin in this group of patients
* Assess significant toxicities in this group of patients and compare to a non-elderly population.
* To determine which clinical parameters will predict lack of completion of six cycles of carboplatin and paclitaxel chemotherapy.
* Assess quality of life changes during chemotherapy and up to one year after completion of chemotherapy.
* Assess progression-free survival and overall survival for this group.
* To determine the feasibility of accrual.

STATISTICAL DESIGN:

Using a one sample binomial design, with 37 patients there was 83% power to detect a null hypothesis of a 45% therapy completion rate versus an alternative hypothesis of a 66% rate assuming a one-sided 5% alpha. The regimen would be declared ineffective if there were 19 or fewer patients who completed 6 cycles of carboplatin and paclitaxel chemotherapy without dose adjustments.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2 and is medically eligible and clinically appropriate to receive systemic chemotherapy
* Diagnosis of ovarian, primary peritoneal, fallopian tube cancer, papillary serous cancer of the endometrium, or mixed mesodermal tumors of the ovary, fallopian tube or uterus
* Life expectancy greater than 6 months
* Baseline laboratory values as described in protocol

Exclusion Criteria:

* Active infection requiring antibiotics at the time of starting chemotherapy
* Prior pelvic radiotherapy > 25% of bone marrow
* Any uncontrolled medical problem that in the opinion of the investigator would preclude safe administration of the study drugs
* Past history of bone marrow transplantation or stem cell support
* Known history of central nervous system (CNS) metastasis
* History of prior malignancy that required prior systemic therapy
* Clinically significant cardiac disease
* Uncontrolled diabetes mellitus
* Any signs of intestinal obstruction
* Participation in an investigational drug study within three weeks prior to study entry
* History of psychiatric disability or other central nervous system disorder

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Matulonis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Matulonis UA, Krag KJ, Krasner CN, Atkinson T, Horowitz NS, Lee H, Penson RT. Phase II prospective study of paclitaxel and carboplatin in older patients with newly diagnosed Mullerian tumors. Gynecol Oncol. 2009 Feb;112(2):394-9. doi: 10.1016/j.ygyno.2008.10.015. Epub 2008 Dec 5. PMID 19058838

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 patients were enrolled between March 26, 2006 and January 2, 2008.
Period: Overall Study
Arm/Group | Carboplatin/Paclitaxel
Started | 12
Completed | 7
Not Completed | 5
Not completed — Death | 2
Not completed — Adverse Event | 1
Not completed — Disease Progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin/Paclitaxel
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 12
Age, Continuous [Mean (Full Range); unit: years] | 78.3 [70 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Therapy Completion Rate
Description: The therapy completion rate is the proportion of patients who completed 6 cycles of carboplatin/paclitaxel therapy without dose reductions.
Time Frame: 6 cycles of therapy, up to approximately 4.5 months given the cycle length of 21 days.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Carboplatin/Paclitaxel
Number analyzed (Participants) | 12
proportion of participants | .50 [0.245 to 0.755]

ADVERSE EVENTS:
Time Frame: The planned treatment regimen was of fixed duration: 6 cycles of therapy, up to approximately 4.5 months given the cycle length of 21 days.
Description: Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAE (v3).
  Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAE (v3).
Groups:
- Carboplatin/Paclitaxel: Paclitaxel: Chemotherapy will be given per standard treatment practices for 6 cycles (18 weeks)
  Carboplatin: Chemotherapy will be given per standard treatment practices for 6 cycles (18 weeks)
Arm/Group | Carboplatin/Paclitaxel
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin/Paclitaxel (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
GI-other (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Infection w/ gr3-4 neut, anal/perianal (Infections and infestations) | 1
Infection-other (Infections and infestations) | 1
Neutrophils (Investigations) | 1
Syncope (Nervous system disorders) | 1
Incontinence urinary (Renal and urinary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin/Paclitaxel (N=12)
Hemoglobin (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Injection site reaction (General disorders) | 1
Pain NOS (General disorders) | 1
Pain-other (General disorders) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 1
Infection-other (Infections and infestations) | 1
Leukocytes (Investigations) | 2
Neutrophils (Investigations) | 2
Platelets (Investigations) | 3
Alkaline phosphatase (Investigations) | 1
ALT, SGPT (Investigations) | 2
AST, SGOT (Investigations) | 1
Creatinine (Investigations) | 1
Metabolic/Laboratory-other (Investigations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 6
Neurologic-other (Nervous system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This study terminated early due to 3 deaths on study and consequently results are limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No